CLINICAL TRIAL: NCT02787421
Title: Predictive Value of Nasal Dilator Strips for Evaluating Nasal Valve Obstruction as Measured by Post-Operative Rhinoplasty Outcomes
Brief Title: Nasal Dilator Strips for Rhinoplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn - changing study design.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Anita Sethna, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00086968
Record Dates: First submitted 2016-05-20; First posted 2016-06-01 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Nasal Valve Compromise
Keywords: Reconstructive Surgery; Rhinoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Rhinoplasty (Experimental): Participants undergoing functional rhinoplasty for nasal valve compromise and obstruction at the Emory Aesthetics Center.
  Interventions: Device: Breathe-Rite Nasal Dilator Strip

INTERVENTIONS:
Device: Breathe-Rite Nasal Dilator Strip — During the pre-operative clinic visit, participants will be given a Breathe-Rite Nasal Dilator Strip

SUMMARY:
In this study, the study team will investigate the validity and role of nasal dilator strips (NDS), a novel method to determine the site of nasal valve compromise (NVC), in the pre-operative evaluation. The method involves placing the strip sequentially at the upper and lower lateral cartilage and recording the location of the optimal airway based on patient's subjective symptoms.

Investigators seek to assess surgical outcomes in participants undergoing rhinoplasty based on pre-operative NDS classification. The Nasal Obstruction and Septoplasty Effectiveness (NOSE) instrument will be used to evaluate subjective symptoms of nasal obstruction, before and after the operation and comparing these scores.The results will help determine the effectiveness and predictive value of NDS in isolating the site of NVC.

DETAILED DESCRIPTION:
In this study, the study team will investigate the validity and role of nasal dilator strips (NDS), a novel method to determine the site of nasal valve compromise (NVC), in the pre-operative evaluation. The method involves placing the strip sequentially at the upper and lower lateral cartilage and recording the location of the optimal airway based on patient's subjective symptoms.

Investigators seek to assess surgical outcomes in participants undergoing rhinoplasty based on pre-operative NDS classification. The Nasal Obstruction and Septoplasty Effectiveness (NOSE) instrument will be used to evaluate subjective symptoms of nasal obstruction, before and after the operation and comparing these scores.The results will help determine the effectiveness and predictive value of NDS in isolating the site of NVC.

Additional study aims are to determine the specificity and predictive value of nasal dilator strips in determining the location of obstruction in patients with nasal valve compromise, and to assess the role of nasal dilator strips in supplementing or replacing current approaches for pre-operative evaluation of nasal valve compromise.

The target population for this study is patients at the Emory Aesthetics Center who are undergoing functional rhinoplasty for nasal valve compromise and obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing functional rhinoplasty for nasal valve compromise and obstruction at the Emory Aesthetics Center

Exclusion Criteria:

* Inability to speak English
* Any disabilities that might prevent patients from completing a survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in Nasal Obstruction and Septoplasty Effectiveness (NOSE) Instrument Score | Prior to surgery and again at 6-10 weeks after surgery
  The NOSE instrument is a highly sensitive assessment of nasal obstruction using participant-reported subjective symptoms. The highest possible score is 100. A higher score indicates more severe nasal congestion symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Sethna, MD, Principal Investigator — Emory University
Locations (1):
- Emory Aesthetic Center, Atlanta, Georgia, United States